CLINICAL TRIAL: NCT01560949
Title: A Phase II Study of Preoperative Systemic Chemotherapy (Modified FOLFIRINOX) Followed by Radiation Therapy for Patients With High Risk Resectable and Borderline Resectable Adenocarcinoma of the Pancreas
Brief Title: Preoperative Folfirinox, Radiation Therapy for Resectable Adenocarcinoma of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1208; NCI-2012-00571 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Adenocarcinoma of the Pancreas; High Risk Resectable; Borderline Resectable; Chemotherapy; Chemoradiation therapy; Oxaliplatin; Eloxatin; Irinotecan; CPT-11; Camptosar; 5-FU; 5-Fluorouracil; Adrucil; Efudex; Gemcitabine; Gemcitabine Hydrochloride; Gemzar; Radiation Therapy; XRT; RT; External Beam Radiation Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Fluorouracil; Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chemotherapy + Radiation (Experimental): SYSTEMIC PHASE: Chemotherapy with Oxaliplatin followed by Irinotecan followed by 5-FU. m FOLFIRINOX - oxaliplatin 75 mg/m2 d1 + irinotecan 150 mg/m2 d1 + 5-FUl 2,000 mg/m2 46h continuous infusion, every other week for 6 cycles (12 weeks).
  CHEMORADIATION PHASE: This phase will start at least 2 weeks, but no more than 6 weeks after completion of the last cycle of mFOLFIRINOX. Chemoradiation with Gemcitabine: 350 mg/m2 IV over 35 minutes every week for 5 doses beginning day 1 (days 1, 8, 15, 22, 29)
  Radiation: External beam radiation therapy will be delivered 5 days/week +/- 2 days over 5.5 weeks with 18-MeV photons. 3D conformal RT, a total dose of 50.4 Gy prescribed to the 95% isodose at 1.8 Gy/fraction (28 fractions) to the GTV + 1.5 cm margin.
  SURGERY- At least 4-6 weeks after last dose of Gemcitabine, if no local progression or distant metastasis. Patients whose scans show unequivocal local or distant progression are not candidates for surgery.
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: 5-FU; Drug: Gemcitabine; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Oxaliplatin — 75 mg/m2 by vein on Day 1 of weeks 1, 3, 5, 7, 9 and 11 for 12 weeks.
  Other Names: Eloxatin
Drug: Irinotecan — 150 mg/m2 by vein on Day 1 of weeks 1, 3, 5, 7, 9 and 11 for 12 weeks.
  Other Names: CPT-11; Camptosar
Drug: 5-FU — 2000 mg/m2 by vein over 46 hour continuous infusion, on Days 1 - 2 during weeks 1, 3, 5, 7, 9 and 11 for 12 weeks.
  Other Names: 5-Fluorouracil; Adrucil; Efudex
Drug: Gemcitabine — 350 mg/m2 by vein every week for 5 doses beginning Day 1 (days 1, 8, 15, 22, 29).
  Other Names: Gemcitabine Hydrochloride; Gemzar
Radiation: Radiation Therapy — External beam radiation therapy delivered 5 days/week +/- 2 days over 5.5 weeks with 18-MeV photons. 3D conformal RT, a total dose of 50.4 Gy 1.8 Gy/fraction (28 fractions).
  Other Names: XRT; RT

SUMMARY:
The goal of this clinical research study is to learn if a chemotherapy combination called modified Folfirinox (or mFolfirinox), followed by a combination of gemcitabine and radiation therapy, followed by surgery, can help to control pancreatic cancer. The safety of this treatment will also be studied.

mFolfirinox consists of 5-FU, oxaliplatin, and irinotecan. These 3 drugs, along with gemcitabine, are each designed to block the growth of cancer cells, which may lead to cancer cell death.

DETAILED DESCRIPTION:
Study Drug Administration:

You will receive up to 3 phases of study therapy: the systemic chemotherapy phase, the chemoradiation phase, and surgery, if possible.

During the systemic chemotherapy phase, you will receive mFolfirinox 1 time every 2 weeks (Weeks 1, 3, 5, 7, 9 and 11) for 12 weeks. You will receive oxaliplatin by vein over a 2-hour period. After receiving oxaliplatin, you will receive irinotecan by vein over a 90-minute period. After receiving irinotecan, you will then receive 5-FU through a portable pump for the next 46 hours. You will take the portable pump home with you and will receive instructions on how to use it.

You will begin receiving chemoradiation within 6 weeks after you have finished receiving the Week 11 dose of mFolfirinox. However, you will not begin receiving it until you have recovered from side effects of the chemotherapy.

During the chemoradiation phase, you will receive gemcitabine over about 35 minutes 1 time each week for 5 weeks. You will also receive radiation therapy 5 days a week (Monday through Friday) for 5 1/2 weeks (a total of 28 treatments). If you miss any of the days of radiation, they will be made up at the end of treatment so that you will receive the full amount of radiation. You will be given a separate consent form that explains the radiation procedure and the risks it may present.

After the chemoradiation phase, you will not receive any treatment for 4-6 weeks so your body can recover. If after this time the disease has not gotten worse or spread to other parts of the body, you will have surgery to try to remove the tumor. You will be given a separate consent form for the surgery that describes how it is performed and its risks.

If the disease has gotten worse or spread to other parts of the body, you will not be able to have surgery. The study doctor will discuss other therapy options with you.

Study Visits:

At Weeks 1, 3, 5, 7, 9, and 11 of the systemic chemotherapy phase:

* You will have a physical exam, including measurement of your weight and vital signs (blood pressure and heart rate).
* Blood (about 3 tablespoons) will be drawn for routine tests.

Within 4 weeks before beginning the chemoradiation phase:

* You will have CT or MRI scans to check the status of the disease.
* Blood (about 1 tablespoon) will be drawn for tumor marker testing.

At Weeks 1, 2, 3, 4, 5, and 6 of the chemoradiation phase:

* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 2-3 tablespoons) will be collected for routine tests. At Week 6, an additional 2 teaspoons of blood will be drawn for CTC testing.

About 4 to 6 weeks after you complete the chemoradiation phase:

* Blood (about 1 tablespoon) will be drawn for tumor marker testing.
* You will have CT or MRI scans to check the status of the disease.

If you are eligible to have surgery after the chemoradiation phase, the following tests and procedures will also be performed:

* Blood (about 4 teaspoons total) will be drawn within 2 weeks before surgery for CTC testing. Blood will also be collected during surgery, if the surgeon thinks it is safe and feasible.
* Tumor tissue collected during a previous procedure will be used for biomarker testing. An additional sample of tumor tissue will be collected from the tissue removed during surgery and used for biomarker testing. Biomarkers are found in the blood/tissue and may be related to your reaction to the study drug.

Length of Study:

You will receive study treatment over the course of up to 30 weeks. You will be taken off study if the disease gets worse, the study doctor thinks it is in your best interest, or if you do not follow the study directions.

You may choose to stop receiving the study treatment at any time. If you choose to stop, you should tell the study doctor or a member of the staff right away. They will make sure that proper procedures are followed and a final visit will be scheduled for your safety.

Follow-up:

Blood (about 2 teaspoons) will be collected for CTC testing 2-3 months after your surgery, if you were one of the first 30 participants enrolled in the study.

You will have a CT or MRI scan of the abdomen and pelvis every 4 months for 2 years to check the status of the disease.

This is an investigational study. 5-FU, oxaliplatin, irinotecan, and gemcitabine are each FDA approved and commercially available to treat different types of cancer:

* 5-FU: pancreatic, gastric, breast, colon/rectum, and skin cancer (basal cell carcinoma)
* Oxaliplatin: colon and rectal cancer
* Irinotecan: colorectal cancer
* Gemcitabine: pancreatic, lung, ovarian, and breast cancer.

The use of these 4 drugs together and in combination with radiation therapy for the treatment of pancreatic cancer is investigational.

Up to 33 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologic or histologic proof of adenocarcinoma of the pancreas is required prior to treatment. Patients with Islet cell tumors are not eligible.
2. Only untreated patients with high risk pancreatic adenocarcinomas will be eligible for the study. For this study, such patients are defined as those who meet one or more of the following radiographic or serologic criteria: a)Primary tumor that involves the superior mesenteric vein causing a vein deformity or segmental venous occlusion with a patent vessel above and below suitable for reconstruction. b)Primary tumor that involves </= 180 degrees of the superior mesenteric artery (SMA), celiac axis or any of its branches on CT or MRI. c) Primary tumor that abuts or encases (>/= 50% of the vessel circumference) a short segment of the common hepatic artery (typically at the gastroduodenal artery origin)
3. (continuation of #2). d) Patients with a high CA19-9 (=/>500mg/dl) in the presence of a bilirubin =/< 2.0 mg/dL. e) Radiographic findings consistent with malignant peripancreatic lymphadenopathy outside the planned field on CT or MRI f) Radiographic findings of indeterminate liver or peritoneal lesions on CT or MRI concerning but not diagnostic of metastatic disease.
4. Patients cannot have known hepatic or peritoneal metastases detected by ultrasound (US), CT scan, MRI or laparotomy.
5. There will be no upper age restriction; patients with Eastern Cooperative Oncology Group (ECOG) 0-1 are eligible.
6. Adequate renal, and bone marrow function: a) Leukocytes >/= 3,000/uL. b) Absolute neutrophil count >/=1,500/uL.c) Platelets >/=100,000/Ul. d) Serum creatinine </= 2.0 mg/dL.
7. Hepatic function (endoscopic or percutaneous drainage as needed). a)Total bilirubin </= 2 X institutional upper limits of normal (ULN). b) AST (SGOT)/ALT (SGPT) </= 5 X institutional ULN.
8. Patients must have no fever or evidence of infection or other coexisting medical condition that would preclude protocol therapy.
9. Women of childbearing potential (defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to practice adequate contraception and to refrain from breast feeding.
10. Patients must sign a study-specific consent form.

Exclusion Criteria:

1. Patients whose tumors are defined as locally advanced cancer or metastatic cancer are not eligible.
2. Unstable angina or New York Heart Association (NYHA) Grade II or greater congestive heart failure; multiple comorbidity that preclude a major abdominal surgery.
3. Known presence of metastases.
4. Inability to comply with study and/or follow-up procedures.
5. Patients < 18 years of age.
6. Pregnant women with a positive (blood B-HCG) pregnancy test are excluded from this study.
7. Patients with an active second malignancy with the exception of non-melanoma skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-06-14 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gauri Varadhachary, MD, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: June 2012 to November 2015. All recruitment done at The University of Texas, MD Anderson Cancer Center.
Pre-assignment Details: A total of 34 participants enrolled in study 1 participant withdrew consent before initiating treatment.
Groups:
- Systemic Phase: mFOLFIRINOX: Systemic: Oxaliplatin at 75 mg/m2 IV on day 1, Irinotecan at 150 mg/m2 IV on day 1, 5 fluorouracil at 2000 mg/m2 IV 46 hour continuous infusion on day 1 - 2, every other week for 6 cycles (12 weeks).
  Chemo: Gemcitabine at 350 mg/m2 IV weekly for 5 doses beginning day 1. External beam radiation therapy delivered 5 days/week, a total dose of 50.4 Gy.
  Surgery: At least 4 - 6 weeks after the last dose of Gemcitabine if there is no local progression or distant metastasis
Period: Systemic Phase: mFOLFIRINOX
Arm/Group | Systemic Phase: mFOLFIRINOX
Started | 33
Completed | 27
Not Completed | 6
Not completed — Adverse Event | 6
Period: Chemoradiation Phase: With Gemcitabine
Arm/Group | Systemic Phase: mFOLFIRINOX
Started | 23
Completed | 23
Not Completed | 0
Period: Surgery Phase
Arm/Group | Systemic Phase: mFOLFIRINOX
Started | 18
Completed | 15
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: A total of 34 participants enrolled in study 1 participant withdrew consent prior to receiving treatment.
Groups:
- Systemic Phase: mFOLFIRINOX: Oxaliplatin at 75 mg/m2 IV on day 1, Irinotecan at 150 mg/m2 IV on day 1, 5 fluorouracil at 2000 mg/m2 IV 46 hour continuous infusion on day 1 - 2, every other week for 6 cycles (12 weeks)
Arm/Group | Systemic Phase: mFOLFIRINOX
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 26
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Resectability Rate
Description: Patients with borderline resectable treated with preoperative modified FOLFIRINOX chemotherapy, followed by gemcitabine-based chemoradiation therapy. At least 4- 6 weeks after the last dose of gemcitabine if there is no local progression or distant metastasis, patients were scheduled for surgery.
Time Frame: 43 months
Measure: Count of Participants; unit: Participants
Groups:
- Surgery: At least 4 - 6 weeks after the last dose of Gemcitabine if there is no local progression or distant metastasis.
Arm/Group | Surgery
Number analyzed (Participants) | 33
Participants | 15

2. Secondary Outcome: Number of Participants With R0 Margin Resection
Description: The specimen was designated R0 if no tumor cells were identified at any of the resection margins.
Time Frame: 43 months
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery
Number analyzed (Participants) | 15
Participants | 10

3. Secondary Outcome: Disease Free Survival (DFS)
Description: Disease free survival (DFS) was defined as the time interval from the date of surgery to the date of disease recurrence or death or the date of a participant was last known to be alive without disease recurrence.
Time Frame: 54 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Phases: Oxalipaltin + irinotecan + 5-fluorouracil, every other week for 6 cycles (12 weeks) followed by gemcitabine weekly for 5 doses with radiation therapy 5 days/week. Then surgery at least 4-6 weeks after the last dose of gemcitabine if no local progression or distant metastasis.
Arm/Group | All Phases
Number analyzed (Participants) | 33
months | 11.1 [5.8 to NA] — Insufficient number of participants with events.

4. Secondary Outcome: Number of Participants That Were SMAD4 Positive Before and After Surgery
Description: Tumor tissue collected pre-therapy and post-therapy for surgically resected patients was assessed for SMAD4 status and classified as either present or absent based on immunohistochemistry evaluation.
Time Frame: 43 months
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery
Number analyzed (Participants) | 15
Participants
  SMAD4 positive before surgery | 4
  SMAD4 positive after surgery | 4

5. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time interval from the date of diagnosis to the date of death due to any cause or the date a patient was last known to be alive. Estimated by using the Kaplan-Meier method.
Time Frame: 54 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Phases(Systematic,Chemoradiation w/ Gemcitabine & Surgery): Oxalipaltin + irinotecan + 5-fluorouracil, every other week for 6 cycles (12 weeks) followed by gemcitabine weekly for 5 doses with radiation therapy 5 days/week. Then surgery at least 4-6 weeks after the last dose of gemcitabine if no local progression or distant metastasis.
Arm/Group | All Phases(Systematic,Chemoradiation w/ Gemcitabine & Surgery)
Number analyzed (Participants) | 33
months | 24 [16.2 to 29.6]

6. Secondary Outcome: Number of Participants With Local and Distant Failure
Time Frame: 43 months
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery
Number analyzed (Participants) | 15
Participants
  Local recurrence | 0
  Distant recurrence | 10

7. Secondary Outcome: Number of Participants Correlative Studies Including DPC4 (SMAD4) Staining and Circulating Tumor Cells (CTC) Pre-Surgery
Description: as for outcome 4
Time Frame: 43 months
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery
Number analyzed (Participants) | 6
Participants
  Present | 4
  Absent | 2

8. Secondary Outcome: Number of Participants Correlative Studies Including DPC4 (SMAD4) Staining and Circulating Tumor Cells (CTC) Post-Surgery
Description: as for outcome 4
Time Frame: 43 months
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery
Number analyzed (Participants) | 11
Participants
  Present | 4
  Absent | 7

ADVERSE EVENTS:
Time Frame: 4 years,6 months
Description: Toxicity was continuously monitored throughout the study, which includes grade 4 hematological toxicity and grade 3 or higher non-hematological toxicity.
Groups:
- Systemin Phase: mFOLFIRINOX: Oxalipaltin 75 mg/m2 IV on day 1, irinotecan 150 mg/m2 IV on day 1, 5-fluorouracil 2,000 mg/m2 IV 46 hours continuous infusion, every other week for 6 cycles (12 weeks).
- Chemoradiation Phase: Radiation With Gemcitabine: Gemcitabine 350 mg/m2 IV weekly for 5 doses beginning day 1. External beam radiation therapy 5 days/week, a total dose of 50.4 Gy.
- Surgery: At least 4-6 weeks after the last dose of gemcitabine if there is no local progression or distant metastasis
Arm/Group | Systemin Phase: mFOLFIRINOX | Chemoradiation Phase: Radiation With Gemcitabine | Surgery
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/23 | 0/18
Serious Adverse Events (participants affected / at risk) | 5/33 | 2/23 | 0/18
Other Adverse Events (participants affected / at risk) | 33/33 | 23/23 | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Systemin Phase: mFOLFIRINOX (N=33) | Chemoradiation Phase: Radiation With Gemcitabine (N=23) | Surgery (N=18)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Gastro-esophageal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Multi-organ failure (Septic shock) (General disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Divice related infection (Infections and infestations) | 1 | 0 | 0
Miocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Atrial fibrilation (Cardiac disorders) | 1 | 0 | 0
Lower respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Systemin Phase: mFOLFIRINOX (N=33) | Chemoradiation Phase: Radiation With Gemcitabine (N=23) | Surgery (N=18)
Diarrhea (Gastrointestinal disorders) | 20 | 5 | 0
Mucositis oral (Gastrointestinal disorders) | 8 | 2 | 0
Vomiting (Gastrointestinal disorders) | 11 | 8 | 0
Fatigue (General disorders) | 28 | 18 | 1
Alanine aminotransferase increased (Investigations) | 13 | 4 | 0
Aspartate aminotranferase increased (Investigations) | 9 | 1 | 0
Alkaline Phosphatase increased (Investigations) | 8 | 4 | 0
Neutrophil count decreased (Investigations) | 10 | 10 | 0
Weight loss (Investigations) | 8 | 5 | 3
Paresthesia (Nervous system disorders) | 13 | 2 | 0
Dysesthesia (Nervous system disorders) | 18 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 11 | 1 | 0
Nausea (Gastrointestinal disorders) | 25 | 15 | 0
Anorexia (Gastrointestinal disorders) | 18 | 10 | 1
Flatulence (Gastrointestinal disorders) | 4 | 2 | 0
Abdominal cramping/pain (Gastrointestinal disorders) | 13 | 7 | 0
Constipation (Gastrointestinal disorders) | 6 | 5 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 9 | 7 | 1
Platelet count (Investigations) | 11 | 18 | 0
Anemia (Blood and lymphatic system disorders) | 7 | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 6 | 0 | 1
Alopesia (Skin and subcutaneous tissue disorders) | 12 | 3 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Flushing (Vascular disorders) | 3 | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Dysguesia (Nervous system disorders) | 5 | 0 | 0
Hyponalbuminemia (Metabolism and nutrition disorders) | 5 | 4 | 0
Musculo-skeletal - other (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-03-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT01560949/Prot_SAP_000.pdf